CLINICAL TRIAL: NCT01133366
Title: A Drug-Drug Interaction Study to Assess the Effects of Multiple Doses of Mipomersen (200 mg SC) on Single-Dose Warfarin (25 mg) Pharmacodynamics and Pharmacokinetics in Healthy Adult Subjects
Brief Title: A Study to Determine the Effects of Multiple Doses of Mipomersen (200 mg SC) on the Pharmacodynamics and Pharmacokinetics of Single-dose Warfarin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kastle Therapeutics, LLC (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MIPO2900509
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
Keywords: ISIS301012; antisense; ApoB (Apolipoprotein B); LDL (low density lipoprotein); mipomersen
MeSH Terms: interventions — Warfarin; mipomersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- warfarin alone (Active Comparator)
  Interventions: Drug: warfarin sodium
- warfarin with mipomersen (Experimental)
  Interventions: Drug: mipomersen sodium; warfarin sodium

INTERVENTIONS:
Drug: warfarin sodium — 25 mg of warfarin oral (single dose)
  Other Names: Coumadin®
  Arms: warfarin alone
Drug: mipomersen sodium; warfarin sodium — 200 mg of mipomersen subcutaneous (SC) (4 doses) plus a single 25 mg of warfarin oral administered with the final mipomersen SC dose
  Other Names: Coumadin®
  Arms: warfarin with mipomersen

SUMMARY:
The purpose of this study is to assess how blood clotting and thinning time is effected when a single dose of warfarin is given alone and when a single dose of warfarin is given with mipomersen; to assess the blood levels of a single dose of warfarin, a single dose of mipomersen, and a single dose of warfarin when given with mipomersen; and to assess the safety of mipomersen when given with or without warfarin.

DETAILED DESCRIPTION:
This will be a Phase 1, open-label, single-sequence, 2-period, crossover study to determine the effect of multiple doses of mipomersen (200 mg SC given every other day for a total of 4 doses) on the PD and PK of warfarin and to evaluate the PK of mipomersen when administered alone and in combination with warfarin. Subjects will be admitted to the clinic on Day -1 until discharge from the clinic on Day 18 and return for outpatient visits on Days 19, 20, and 78. All subjects will receive a single 25-mg oral dose of warfarin given alone on Day 1 (designated the reference treatment). All subjects will then receive 200-mg SC doses of mipomersen given every other day on Days 8, 10, 12, and 14 (total of 800 mg mipomersen) with a single 25-mg oral dose of warfarin also given on Day 14 (combination designated the test treatment).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent before any study-related procedure is performed.
* Body mass index (BMI) between 18 and 32 kg/m2, inclusive.
* No clinically significant abnormalities based on medical history, laboratory assessments, vital sign, 12-lead electrocardiogram (ECG) results, and physical examination.
* Subjects willing and able to follow a prescribed diet.
* Subjects have not consumed nicotine or nicotine-containing products for at least 6 months before Screening.
* Subjects are nonpregnant and nonlactating, surgically sterile, postmenopausal, abstinent, or the subject or partner is willing to use a reliable method of contraception during the study and for 5 months after mipomersen dosing.

Exclusion Criteria:

* Poor metabolizer of warfarin as determined by CYP2C9 genotype testing.
* Clinically significant PT, aPTT, INR, protein C, protein S, or platelet count results or hematuria.
* Abnormal prolongation of skin bleeding time or a personal or family history of coagulation or bleeding disorders, vascular malformations including aneurysms, or venous thromboembolism.
* Active or recurring clinically significant cardiovascular, pulmonary, renal, endocrine, hepatic, neurologic, psychiatric, immunologic, hematologic, gastrointestinal, or metabolic disease.
* Active malignancy of any type other than nonmelanomatous skin malignancies.
* Use of any prescribed or over-the-counter concomitant medications within 14 days before the first dose of investigational product without approval of the Investigator and Sponsor.
* Positive test result for drugs of abuse, alcohol, or cotinine or history of alcohol abuse or drug addiction.
* Positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or HIV.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-05; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Area under the effect curve (AUC), for INR (international normalized ratio), PT (prothrombin time), and aPTT (activated partial thromboplastin time) | Serial sampling up to 144 hours post dose
Maximal Value (MAX) for INR, PT and aPTT | Serial sampling up to 144 hours post dose
Time of maximal effect (Tmax) for INR, PT, and aPTT | Serial sampling up to 144 hours post dose

SECONDARY OUTCOMES:
Warfarin Plasma Pharmacokinetic parameters (AUC 0-t, AUC 0-inf, Maximum Concentration (Cmax)) | Serial PK sampling up to 144 hours post dose
Mipomersen Plasma Pharmacokinetic parameters (AUC0-t, AUC0-inf, Cmax) | Serial PK sampling up to 24 hours post dose
Incidence of treatment-emergent Adverse Events | Through Day 78

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- PPD Development, LP, Austin, Texas, United States